CLINICAL TRIAL: NCT01559740
Title: Transversus Abdominis Plane Blocks for Infants and Children for Postoperative Pain Control: Is it the Concentration or Volume of Local Anesthetic Solution That Improves Analgesia?
Brief Title: Transversus Abdominis Plane Blocks for Infants and Children for Postoperative Pain Control
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CMH IRB 2009-13887
Record Dates: First submitted 2012-03-12; First posted 2012-03-21 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Postoperative Pain
Keywords: regional anesthesia; children; postoperative pain relief
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.25% Bupivacaine (Experimental): All children will receive a single dose of 1 mcg/kg of Fentanyl intravenously prior to incision. Group TAP 1 receiving a TAP block with 0.25% bupivacaine with 1:200,000 epinephrine at a dose of 1 mL/kg.
  Interventions: Drug: Bupivacaine
- 0.125% Bupivacaine (Experimental): All children will receive a single dose of 1 mcg/kg of Fentanyl intravenously prior to incision. Group TAP 2 will receive a TAP block with a total dose of 1 mL/kg given at a concentration of 0.125% bupivacaine with 1:200,000 epinephrine.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — This is being used as the local anesthetic for the TAP blocks at either 0.25% or 0.125%. The block will be done once during the procedure.

SUMMARY:
After undergoing hernia surgery, hydrocelectomy or lower abdominal surgery, a child may experience some amount of pain in the post-operative period. As part of the anesthesia technique, the investigators routinely provide a nerve block done on the abdominal wall that will provide pain relief for at least 10 hours postoperatively. This is referred to as a TAP block. The purpose of this study is to determine if the nerve block performed with local anesthetic solution using a regular concentration solution vs. a diluted solution may offer different durations of pain relief.

DETAILED DESCRIPTION:
Children undergoing groin surgery or abdominal surgery under general anesthesia are offered pain relief postoperatively using regional anesthesia techniques including a central block like a caudal block, or peripheral nerve blocks including ultrasound guided ilioinguinal nerve block or transversus abdominis plane (TAP) block. The TAP block, a peripheral block of the thoraco-lumbar nerve roots as they exit between the internal oblique and the transversus abdominis muscle can be easily visualized using ultrasound guidance. The TAP block has been used for analgesia following major surgeries including lower abdominal surgeries and in newborn infants following major abdominal procedures including colostomy placement.1 The purpose of this study is to determine if two different concentrations of bupivacaine delivered at a total dose of 1 mL/kg offer similar or altered analgesia, i.e., does the concentration of the anesthetic matter more than the volume of local anesthetic while performing a TAP block in children undergoing groin surgery. Parents and the investigators will be blinded to the solution used for the TAP block. The solution will be drawn up by an investigator who is not a participant in the patient's care in a sterile fashion.

ELIGIBILITY:
Inclusion Criteria:

* Children under 8 years of age presenting for hernia repair, hydrocelectomy or lower abdominal surgery
* Estimated operative time approximately 3 hours
* American Society of Anesthesiologists Classification ASA I or II
* Parental consent to be included in the study

Exclusion Criteria:

* Any contraindications to local anesthesia but not limited to

  1. Local infection of the abdominal wall.
  2. Allergy to amide local anesthetics
  3. History of significant cardiac disease or uncontrolled seizures.
  4. Allergy to rescue analgesia including acetaminophen and or hydromorphone.
  5. Neonates under 28 days.
* Inability for the family to complete the postoperative questionnaire

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
TAP Block Concentration of Bupivacaine that Reduces Postoperative Pain | Participants will be followed for the duration of anesthesia and after surgery, an average of 48 hours
  The difference in concentrations will be measured by using FLACC score every 5 mins for one hour after surgery in the Post Anesthesia Care Unit. Blood pressuer and heart rate will also be recorded.

SECONDARY OUTCOMES:
Dose of rescue medications given between the two groups | Participants will be followed for the duration of anesthesia and after surgery, an average of 48 hours
  The dose of pain medications administered will be recorded by the nurse or study coordinator while in the hospital. The caregiver will record the dose of pain medications administered in a caregiver questionnaire sheet.
Number of rescue medications given between the two groups | Participants will be followed for the duration of anesthesia and after surgery, an average of 48 hours
  The number of pain medications administered will be recorded by the nurse or study coordinator while in the hospital. The caregiver will record the number of pain medications administered in a caregiver questionnaire sheet.
Time the rescue medications were administered between the two groups | Participants will be followed for the duration of anesthesia and after surgery, an average of 48 hours
  The time pain medications administered will be recorded by the nurse or study coordinator while in the hospital. The caregiver will record the time pain medications administered in a caregiver questionnaire sheet.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Bielsky A, Efrat R, Suresh S. Postoperative analgesia in neonates after major abdominal surgery: 'TAP' our way to success! Paediatr Anaesth. 2009 May;19(5):541-2. doi: 10.1111/j.1460-9592.2009.02988.x. No abstract available. PMID 19453587
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Suresh S, Chan VW. Ultrasound guided transversus abdominis plane block in infants, children and adolescents: a simple procedural guidance for their performance. Paediatr Anaesth. 2009 Apr;19(4):296-9. doi: 10.1111/j.1460-9592.2009.02958.x. PMID 19335342